CLINICAL TRIAL: NCT00809224
Title: Tracking Brain Changes During Real and Imagined Movements in People With ALS (Lou Gehrig's Disease) and Healthy Volunteers.
Brief Title: Cortex Changes in Real/Imagined Movements in Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Robert Welsh, Research Associate Professor, University of Michigan
Other Study IDs: R01NS052514 (NIH); Hum00000219
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: ALS; Amyotrophic Lateral Sclerosis
Keywords: ALS; amyotrophic lateral sclerosis; brain-computer interface; functional magnetic resonance imaging; radiology; fMRI
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ALS: ALS group should have ALS.
- Control: The control group should not have ALS or any other neurological/psychiatric disorder, and must be over the age of 40.

SUMMARY:
The purpose of this study is to track areas of the brain, via functional magnetic resonance imaging (fMRI), that retain structural and functional integrity throughout the lifespan of people with amyotrophic lateral sclerosis (ALS), also known as Lou Gehrig's disease.

DETAILED DESCRIPTION:
A severe physical disability has a dramatic impact on a person's life, whether it is caused by a neuro-degenerative disease such as amyotrophic lateral sclerosis (ALS), a brainstem stroke, or a spinal cord injury. Someone with these conditions may be effectively "locked-in," retaining their cognitive ability, but unable to perform any movement except, possibly, the most basic eye movements.

Areas of the brain that retain structural and functional integrity throughout the lifespan of people with ALS may be suitable for a technology called brain-computer interfaces (BCI). One day, BCIs-which can be operated "just by thinking"-may allow people with neurological disorders, such as ALS, to communicate and regain some mobility with the assistance of electronic devices.

In this study we will use functional magnetic resonance imaging (fMRI) to track areas of the brain that retain structural and functional integrity throughout the lifespan of people with ALS.

The trial involves visits to the study facility every 2-6 months for up to 30 months or until visits are no longer possible. During each visit, participants will undergo a fMRI exam. During that time they will view visual images and be asked to perform 4 different motor tasks: 1) actual finger tapping, 2) actual fist clenching, 3) imaginary finger tapping, and 4) imaginary fist clenching. Each of the mini-experiments (tasks) lasts for about 6-7 minutes. While the participants are performing the tasks their brains will be repeatedly imaged using fMRI. We will then use the images to look for correlations to the tasks, which in turn will result in identifying the brain areas responsible for the activities. After the fMRI, participants will be asked to fill out questionnaires. Performing the tasks takes about 90 minutes and filling out the questionnaires takes about 30 minutes.

The facility is located on the North Campus of the University of Michigan-Ann Arbor. The study coordinators currently are enrolling participants with ALS and creating a database of healthy volunteers whom they will contact at a later date.

Information gained from this study will contribute to a better understanding of ALS disease progression, and could lead to significant quality-of-life improvements for persons with end-stage ALS.

ELIGIBILITY:
Inclusion Criteria:

Participants with and without ALS must:

* be between 18 and 70 years of age
* not be claustrophobic
* not have metal particles in their eyes
* not have metal implants (joints, inner ear, pacemaker, etc.) or foreign metal in their body
* not have a history of neurological or psychiatric disorder
* not have a history of alcohol or drug abuse
* be able to lie on their back for 90 minutes
* not be dependent on artificial ventilation
* not be on PiPap, or must be capable of being off it for greater than 6 hours
* healthy controls must be over the age of 40

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All are able to participate.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2008-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
cortical activation patterns | Yearly

CONTACTS AND LOCATIONS:
Overall Officials: Robert Welsh, PhD, Principal Investigator — Research Assistant Professor, University of Michigan Department of Radiology
Locations (1):
- University of Michigan, Functional MRI Laboratory, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Abrahams S, Goldstein LH, Simmons A, Brammer M, Williams SC, Giampietro V, Leigh PN. Word retrieval in amyotrophic lateral sclerosis: a functional magnetic resonance imaging study. Brain. 2004 Jul;127(Pt 7):1507-17. doi: 10.1093/brain/awh170. Epub 2004 May 26. PMID 15163610
- [Background] Biswal BB, Van Kylen J, Hyde JS. Simultaneous assessment of flow and BOLD signals in resting-state functional connectivity maps. NMR Biomed. 1997 Jun-Aug;10(4-5):165-70. doi: 10.1002/(sici)1099-1492(199706/08)10:4/53.0.co;2-7. PMID 9430343
- [Background] Brooks BR, Bushara K, Khan A, Hershberger J, Wheat JO, Belden D, Henningsen H. Functional magnetic resonance imaging (fMRI) clinical studies in ALS--paradigms, problems and promises. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Jun;1 Suppl 2:S23-32. doi: 10.1080/14660820052415790. PMID 11464937
- [Background] Havel P, Braun B, Rau S, Tonn JC, Fesl G, Bruckmann H, Ilmberger J. Reproducibility of activation in four motor paradigms. An fMRI study. J Neurol. 2006 Apr;253(4):471-6. doi: 10.1007/s00415-005-0028-4. Epub 2005 Nov 14. PMID 16283098
- [Background] Jacob S, Finsterbusch J, Weishaupt JH, Khorram-Sefat D, Frahm J, Ehrenreich H. Diffusion tensor imaging for long-term follow-up of corticospinal tract degeneration in amyotrophic lateral sclerosis. Neuroradiology. 2003 Sep;45(9):598-600. doi: 10.1007/s00234-003-1014-0. Epub 2003 Aug 7. PMID 12904924
- [Background] Konrad C, Henningsen H, Bremer J, Mock B, Deppe M, Buchinger C, Turski P, Knecht S, Brooks B. Pattern of cortical reorganization in amyotrophic lateral sclerosis: a functional magnetic resonance imaging study. Exp Brain Res. 2002 Mar;143(1):51-6. doi: 10.1007/s00221-001-0981-9. Epub 2002 Jan 24. PMID 11907690
- [Background] Konrad C, Jansen A, Henningsen H, Sommer J, Turski PA, Brooks BR, Knecht S. Subcortical reorganization in amyotrophic lateral sclerosis. Exp Brain Res. 2006 Jul;172(3):361-9. doi: 10.1007/s00221-006-0352-7. Epub 2006 Mar 25. PMID 16463149
- [Background] Sach M, Winkler G, Glauche V, Liepert J, Heimbach B, Koch MA, Buchel C, Weiller C. Diffusion tensor MRI of early upper motor neuron involvement in amyotrophic lateral sclerosis. Brain. 2004 Feb;127(Pt 2):340-50. doi: 10.1093/brain/awh041. Epub 2003 Nov 7. PMID 14607785
- [Background] Schoenfeld MA, Tempelmann C, Gaul C, Kuhnel GR, Duzel E, Hopf JM, Feistner H, Zierz S, Heinze HJ, Vielhaber S. Functional motor compensation in amyotrophic lateral sclerosis. J Neurol. 2005 Aug;252(8):944-52. doi: 10.1007/s00415-005-0787-y. Epub 2005 Mar 6. PMID 15750701